CLINICAL TRIAL: NCT06069817
Title: Impact of High Flow Therapy Through Nasal Cannula on Complications Related to Airway Stenting: a Prospective, Multicentric, Randomized-controlled Trial
Brief Title: Impact of High Flow Therapy on Complications Related to Airway Stenting
Acronym: HiSTENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardarelli Hospital (Other)
Responsible Party: Principal Investigator, Giuseppe Failla, Chief of Interventional Pulmonology Unit, Cardarelli Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1A
Record Dates: First submitted 2023-09-25; First posted 2023-10-06 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Airway Obstruction; Respiratory Infection; Mucus; Plug
Keywords: high flow nasal cannula; airway stent; nebulized saline
MeSH Terms: conditions — Airway Obstruction; Respiratory Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal cannula group (Experimental): Treatment with High Flow Nasal Cannula minimum twenty (20) minutes three times a day (one [1] hour a day in total) and up to 10 hours a day in total, according to patient's preferences.
  Interventions: Device: High flow nasal cannula
- nebulized saline group (Active Comparator): Treatment with nebulization of 4-8 cc of normal saline three times daily
  Interventions: Device: nebulized normal saline

INTERVENTIONS:
Device: High flow nasal cannula — home treatment with HFNC after airway stent placement both for malignant and benignant central airway obstruction
  Arms: High flow nasal cannula group
Device: nebulized normal saline — home treatment with nebulized normal saline after airway stent placement both for malignant and benignant central airway obstruction
  Arms: nebulized saline group

SUMMARY:
The application of HFNC therapy in patients with airway stent, improving both humidification and clearance of the airway secretion, could potentially reduce the risk of mucoid impaction, respiratory infections and granulation. HFNC therapy could be superior to nebulization of normal saline (usual care) in order to keep the stent cleaned, reducing, by inference, the risk of complications, as defined above.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Central Airway obstruction, both malignant and nonmalignant, treated with airway stenting (silicone or fully covered metallic stent)

Exclusion Criteria:

* Contraindication to HFNC (recent - within 3 months - nose surgery or facial trauma)
* Lack of written informed consent
* Neuropsychiatric disorders
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of mucous plugging associated with airway stent in HFNC group | within 7 days from stent placement
  mucous plugging assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of mucous plugging associated with airway stent in HFNC group | within 30 days from stent placement
  mucous plugging assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of mucous plugging associated with airway stent in HFNC group | within 60 days from stent placement
  mucous plugging assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of mucous plugging associated with airway stent in HFNC group | within 90 days from stent placement
  mucous plugging assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of mucous plugging associated with airway stent in nebulized saline group | within 7 days from stent placement
  mucous plugging assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of mucous plugging associated with airway stent in nebulized saline group | within 30 days from stent placement
  mucous plugging assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of mucous plugging associated with airway stent in nebulized saline group | within 60 days from stent placement
  mucous plugging assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of granuloma associated with airway stent in HFNC group | within 90 days from stent placement
  granuloma formation assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of granuloma associated with airway stent in nebulized saline group | within 7 days from stent placement
  granuloma formation assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of granuloma associated with airway stent in nebulized saline group | within 30 days from stent placement
  granuloma formation assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of granuloma associated with airway stent in nebulized saline group | within 60 days from stent placement
  granuloma formation assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of granuloma associated with airway stent in nebulized saline group | within 90 days from stent placement
  granuloma formation assessed during bronchoscopy, eventually determining reduction in cross-sectional stent area
incidence of respiratory infection associated with airway stent in HFNC group | within 90 days from stent placement
  symptoms of respiratory infection + radiologic and/or bronchoscopic signs of infection + need of antibiotic therapy
incidence of respiratory infection associated with airway stent in nebulized saline group | within 90 days from stent placement
  symptoms of respiratory infection + radiologic and/or bronchoscopic signs of infection + need of antibiotic therapy

SECONDARY OUTCOMES:
adherence to home treatment with HFNC in patients with airway stent, as assesed by time of daily utilization | within 90 days from stent placement
  minutes a day spent on HFNC
adherence to home treatment with nebulization of normal saline in patients with airway stent, as assesed by time of daily utilization | within 90 days from stent placement
  times a day spent on nebulization
incidence of adverse events due to home treatment with HFNC in patients with airway stent | within 90 days from stent placement
  incidence of malfunction of the device; incidence of complications as assessed by clinical examination (cough, headache, rhinitis)
incidence of adverse events due to home treatment with nebulization of normal saline in patients with airway stent | within 90 days from stent placement
  incidence of malfunction of the device; incidence of complications as assessed by clinical examination (cough, headache, rhinitis)
Satisfaction of home treatment with HFNC by Cough and sputum assessment questionnaire (CASA-Q) | within 90 days from stent placement
  Cough and sputum assessment questionnaire (CASA-Q) to evaluate both severity of cough and sputum production to quality of life impairment (minimum value 0, maximum value 100; higher scores mean worse outcome)
Satisfaction of home treatment with nebulized saline by Cough and sputum assessment questionnaire CASA-Q | within 90 days from stent placement
  Cough and sputum assessment questionnaire (CASA-Q) to evaluate both severity of cough and sputum production to quality of life impairment (minimum value 0, maximum value 100; higher scores mean worse outcome)
incidence of airway stent colonization in HFNC group | within 90 days from stent placement
  positive bronchial aspirate culture
incidence of airway stent colonization in nebulized saline group | within 90 days from stent placement
  positive bronchial aspirate culture
all cause-mortality in HFNC group | within 90 days from stent placement
all cause-mortality in nebulized saline group | within 90 days from stent placement
mortality due to respiratory infection in HFNC group | within 90 days from stent placement
mortality due to respiratory infection in nebulized saline group | within 90 days from stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Failla, MD, Study Director — Ospedale "Antonio Cardarelli", Naples; Nadia Corcione, MD, PhD, Principal Investigator — Ospedale "Antonio Cardarelli", Naples; Alfonso Pecoraro, MD, Principal Investigator — Ospedale "Antonio Cardarelli", Naples
Locations (1):
- Interventional Pulmonology Unit, Cardarelli Hospital, Napoli, Italy